CLINICAL TRIAL: NCT03860532
Title: Phase I Randomized,Double-Blind,Placebo-controlled Trial in Healthy Male Voluteers To Examine the Safety,Tolerability,and Pharmacokinetics of HMPL-011 After A Single Dose.
Brief Title: Phase I Clinical Trial in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2009-011-00AU1
Record Dates: First submitted 2012-03-15; First posted 2019-03-04 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HMPL-011 tablets (Active Comparator): A sigle total oral dose of 1200 mg tablets (600 mg tablet X 2)
  Interventions: Drug: HMPL-011 tablets
- HMPL-011 capsules (Active Comparator): A sigle total oral dose of 1200 mg capsules (200 mg tablet X 6)
  Interventions: Drug: HMPL-011 capsules

INTERVENTIONS:
Drug: HMPL-011 tablets — Eligible subjects will recieve 1200 mg HMPL-011 tablets under fed and diet circumstance.
  Arms: HMPL-011 tablets
Drug: HMPL-011 capsules — Eligible subjects will recieve 1200 mg HMPL-011 capsules under fed and diet circumstance.
  Arms: HMPL-011 capsules

SUMMARY:
This is a Phase I Randomized,Double-Blind,Placebo-controlled Trial in Healthy Male Voluteers To Examine the Safety,Tolerability,and Pharmacokinetics of HMPL-011 After A Single Dose.

DETAILED DESCRIPTION:
Eligible subjects will randomly recieve 1200 mg tablets (600 mg tablet X 2) or 1200 mg capsules (200 mg capsule X 6) of HMPL-011 under fed and fed circumstance in part 1. In part 2, eight subjects will be enrolled and given 800 mg tablets (400 mg/tablet X 2) every 8 hours daily for 6 days (morning dose only on Day 6).

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following criteria at the Screening Visit will be eligible to participate in the study:

* Healthy adult male and female subjects, 18-70 years of age, inclusive, at the time of signing the informed consent;
* Body weight ≥ 50 kg and body mass index (BMI) within the range 19-30 kg/m2, inclusive, at screening;
* Medically healthy subjects with clinically insignificant screening and check-in results (medical histories, 12-lead ECG, physical exam and laboratory tests);
* Female subjects of childbearing potential with a negative urine pregnancy test at screening who are not breastfeeding, do not plan to become pregnant during the study, and agree to use an approved method of birth control from the first dose until 7 days following the last administration of study drug;
* Male subjects must agree to use barrier contraception (condom with spermicide) in addition to having their female partner (if of child-bearing potential) use another acceptable form of contraception (IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, or subdermal hormonal implant) from first dose until 7 days following the last administration of study drug; and
* Subjects are able to understand and to give their signed informed consent before any trial related procedures being performed.

Exclusion Criteria:

Subjects are excluded from participation in the study if any of the following criteria apply:

* Subjects with, or a history of, cancer, diabetes or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, hematological, dermatological, venereal, neurological, psychiatric or other major disorder;
* Presence or history of GI, hepatic or renal disease or any other condition (including surgery) known to interfere with the absorption, distribution, metabolism or excretion of medicines; Hutchison MediPharma Ltd. Clinical Study Protocol HMPL-004-1002 Confidential & Proprietary 27 Final 20 July 2011
* Systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 40 to 90 mmHg, and/or pulse rate outside the range of 40 to 100 bpm after one repeat at screening or check-in;
* Abnormal ECGs at screening
* History of clinically significant drug and/or food allergies as determined by the Principal Investigator (PI);
* Subjects will be excluded if they experience arrhythmia of any clinical significance;
* Subject is not willing to abstain from alcohol for 48 hours prior to the start of the first dose until completion of the post-study follow-up assessments;
* Any history (within 2 years) or current diagnosed alcoholism defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (One unit is equivalent to a half-pint of beer or 1 measure of spirits or 1 glass of wine.);
* Recent history or current diagnosed drug abuse;
* Tobacco or nicotine use within the 6 months prior to first dose until the follow-up assessment, or a positive urine screen for cotinine;
* Hypersensitivity or idiosyncratic reaction to compounds related to the study drug;
* Use of substances known to be strong inhibitors or inducers of cytochrome P450 enzymes (eg, macrolides, calcium channel blockers, ritonavir, rifampin, St. John's Wort, etc.) within 30 days prior to the first dose;
* Use of prescription or non-prescription drugs, including high-dose vitamins, herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication (except for strong inhibitors or inducers of cytochrome P450 enzymes);
* Consumption of food or beverage containing grapefruit or cranberry within 7 days prior to the dose of study medication;
* Recent significant changes in body weight due to dieting or nutritional treatment;
* Donation of whole blood in excess of 500 mL within 56 days prior to checkin;
* Plasma donation within 7 days prior to check-in;
* Subject participated in an investigational clinical study within 30 days prior to the first dosing, or days calculated as ten times the half-life of the compound which the subject was treated with, whichever is longer. Factors other than the half-life of the compound, such as accumulation of tissue, muscle or organ, should also be considered for the enrollment;
* Exposure to 4 or more investigational products within 12 months prior to the first dosing day; Hutchison MediPharma Ltd. Clinical Study Protocol HMPL-004-1002 Confidential & Proprietary 28 Final 20 July 2011
* Positive screen for HIV, hepatitis B, and/or hepatitis C at screening;
* Positive urine screen for drugs of abuse at screening or check-in; and
* Any condition that, in the opinion of the Principal Investigator, would complicate or compromise the study, or the well-being of the subject 4.2.3 General and Dietary Restrictions

The following items are not to be consumed for 48 hours (2 days) prior to the first dose until the last scheduled blood sample collection of the study:

* Caffeine/xanthine such as coffee, tea, chocolate, and all caffeine containing soft drinks or energy drinks;
* Alcoholic beverages and/or other alcohol containing products; and
* Any foods containing poppy seeds.

The following items are not to be consumed for 14 days prior to the first dose and throughout the study until the last scheduled blood sample collection:

• Grapefruit, pomelo, cranberry, or grapefruit, pomelo, or cranberry-containing products. While in the CPU, subjects will not be allowed additional sugar in beverages or on cereal, though limited use of other sweeteners is allowed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of HMPL-011 tablets vs capsules in fasted States | 72 hours
  Peak Plasma Concentration (Cmax) of HMPL-011 tablets (600 mg tablet X 2) and capsules (200 mg capsule X 6) in fasted States.
Peak Plasma Concentration (Cmax) of HMPL-011 tablets vs capsules in fed States | 72 hours
  Peak Plasma Concentration (Cmax) of HMPL-011 tablets (600 mg tablet X 2) and capsules (200 mg capsule X 6) in fed States.
Steady State concentration of HMPL-011 | 5 weeks
  Steady State concentration of HMPL-011 will be caculated based on Ctrough
Area under the plasma concentration versus time curve (AUC) of HMPL-011 tablets vs capsules in fed States. | 72 hours
  Area under the plasma concentration versus time curve (AUC) of HMPL-011 tablets (600 mg tablet X 2) and capsules (200 mg capsule X 6) in fed States.
Area under the plasma concentration versus time curve (AUC) of HMPL-011 tablets vs capsules in fasted States. | 72 hours
  Area under the plasma concentration versus time curve (AUC) of HMPL-011 tablets (600 mg tablet X 2) and capsules (200 mg capsule X 6) in fasted States.

SECONDARY OUTCOMES:
Overall incidence of TEAEs | 5 weeks
  The proportion of subjects reported at least 1 TEAE